CLINICAL TRIAL: NCT07302711
Title: Evaluation of the Effectiveness of Pericapsular Nerve Group Block in Hemiplegic Shoulder Pain
Status: Not yet recruiting | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 09.2025.25-0859
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-11

CONDITIONS: Shoulder Pain; Hemiplegia
Keywords: PENG block; shoulder joint pain; Hemiplegic shoulder
MeSH Terms: conditions — Shoulder Pain; Hemiplegia | interventions — Dental Occlusion

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: All participants will receive a single ultrasound-guided Pericapsular/Periarticular Nerve Group (PENG) block
  Interventions: Procedure: Ultrasound-Guided Pericapsular/Periarticular Nerve Group (PENG) Block

INTERVENTIONS:
Procedure: Ultrasound-Guided Pericapsular/Periarticular Nerve Group (PENG) Block — Under real-time ultrasound guidance, a 100-mm needle is advanced in-plane between the deltoid muscle and the subscapularis tendon with the patient in the supine position and the affected arm externally rotated and abducted at approximately 45 degrees.
  A total of 10 mL of 0.25% bupivacaine hydrochloride combined with 4 mg of dexamethasone is injected slowly into the pericapsular space to provide analgesia to the glenohumeral joint.

SUMMARY:
Hemiplegic shoulder pain (HSP) is a common and clinically significant complication after stroke that negatively affects rehabilitation outcomes. It is associated with shoulder subluxation, capsular contracture, spasticity, and central pain mechanisms, leading to pain, limited range of motion, and reduced quality of life. The suprascapular nerve (SSN) block has been shown to be effective for shoulder pain management; however, the glenohumeral joint (GHJ) receives innervation from multiple nerves including the axillary, subscapular, and lateral pectoral nerves. The recently described pericapsular/periarticular nerve group (PENG) block targets these articular branches and may provide analgesia with minimal motor impairment.

This study aims to evaluate the effects of adding an ultrasound-guided PENG block to conventional physical therapy in patients with post-stroke hemiplegic shoulder pain, focusing on pain intensity, range of motion, and quality of life outcomes.

DETAILED DESCRIPTION:
Pericapsular/Periarticular Nerve Group (PENG) Block Procedure:

The procedure is performed with the patient in the supine position, the affected arm externally rotated and abducted approximately 45 degrees. A high-frequency linear ultrasound probe is placed longitudinally between the coracoid process and the humeral head. After identifying the humeral head, the subscapularis muscle tendon, and the overlying deltoid muscle, an in-plane approach is used to advance a 100-mm needle between the deltoid muscle and the subscapularis tendon under real-time ultrasound guidance.

After confirming the needle tip position, a total of 10 mL of 0.25% bupivacaine hydrochloride combined with 4 mg of dexamethasone is injected slowly, ensuring appropriate spread within the targeted pericapsular space. The goal of the block is to provide analgesia for the glenohumeral joint by targeting the articular branches of the axillary, subscapular, and lateral pectoral nerves with minimal motor impairment.

No major complications have been reported for this technique in the literature. However, minor complications such as local bleeding, infection, or transient vasovagal reactions may occur.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 85 years

Stroke onset less than 1 year

Presence of hemiplegic shoulder pain with limited shoulder range of motion confirmed by clinical examination

Numeric Rating Scale (NRS) pain score ≥ 4

Exclusion Criteria:

* Severe deformity or pathology of the shoulder region

Complex regional pain syndrome type I

Modified Ashworth Scale score ≥ 3

Presence of neglect syndrome

Grade 4 glenohumeral joint degeneration

Coagulopathy or bleeding disorders

Fracture on the affected side

Secondary pathology on MRI (malignancy or infection)

Presence of pacemaker

History of allergic reaction to local anesthetic agents or dexamethasone

Shoulder intervention or injection within the past 3 months

Major psychiatric illness

Refusal to participate in the study

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 to 85 years with post-stroke hemiplegic shoulder pain and limited shoulder joint range of motion will be recruited from the Pain Medicine and Physical Therapy Departments of Marmara University Pendik Training and Research Hospital. All participants will have experienced a stroke within the past year and will present with a Numeric Rating Scale (NRS) pain score of 4 or higher at baseline.
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-03-20 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Intensity (Numeric Rating Scale, NRS): | Baseline, 1 hour, 2 weeks, and 2 months post-intervention. Numeric Rating Scale
  NRS is a scale in which the patient gives points between "0" and "10" for the low back and leg pain felt by the patient, "0" = No pain, "10" = The most severe, unbearable pain

SECONDARY OUTCOMES:
Fugl-Meyer Assessment for Upper Extremity (FMA-UE) | Baseline, 2 weeks, and 2 months
  The Fugl-Meyer Upper Extremity Scale is a validated assessment tool designed to evaluate motor recovery after stroke. It includes motor function of the upper limb, wrist, hand movements, coordination, and reflex activity. Each item is scored from 0 to 2 (0 = cannot perform, 1 = partial performance, 2 = normal performance), with a total possible score of 66 points.
Quick Disabilities of the Arm, Shoulder, and Hand (QuickDASH) Questionnaire | Baseline, 2 weeks, and 2 months
  The QuickDASH is an 11-item self-reported questionnaire measuring upper extremity function and symptoms. Scores range from 0 to 100, where higher scores indicate greater disability.
Modified Ashworth Scale (MAS) | Baseline, 2 weeks, and 2 months
  The MAS is a clinical tool used to assess muscle tone and spasticity. Muscle tone is rated from 0 (no increase in tone) to 4 (rigid in flexion or extension). Higher scores indicate more severe spasticity.
Stroke-Specific Quality of Life Scale (SS-QOL) | Baseline, 2 weeks, and 2 months
  The SS-QOL is a 49-item stroke-specific scale assessing 12 domains related to quality of life, including mobility, upper extremity function, mood, energy, social roles, language, and thinking. Each item is rated on a 5-point Likert scale; higher scores represent better quality of life.
Modified Barthel Index (MBI) | Baseline, 2 weeks, and 2 months
  The MBI assesses activities of daily living (ADL) and functional independence. Scores range from 0 to 100, with higher scores indicating greater independence.
Shoulder Range of Motion (ROM) | Baseline, 2 weeks, and 2 months
  Active and passive shoulder joint range of motion (flexion, abduction, internal and external rotation) will be measured using a goniometer. The range will be recorded at the point of pain onset and maximum movement.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)